CLINICAL TRIAL: NCT02915484
Title: Transcranial Direct Current Stimulation (tDCS) in Chronic Post-Stroke Apathy
Acronym: TDCS-PSA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with recruitment.
Sponsor: Stony Brook University (Other)
Collaborators: National Center of Neuromodulation for Rehabilitation (Other)
Responsible Party: Principal Investigator, Andrew Goldfine, MD, Stony Brook University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 798869
Record Dates: First submitted 2016-09-20; First posted 2016-09-27 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Apathy; Stroke
Keywords: Transcranial Direct Current Stimulation; Apathy; Stroke; Empathy; Electric Stimulation Therapy; Depression; Anhedonia; Prefrontal Cortex; Electroencephalography; Cognition; Emotions; Neurological Rehabilitation; Brain Diseases; Cerebrovascular Disorders
MeSH Terms: conditions — Lethargy; Stroke; Depression; Anhedonia; Brain Diseases; Cerebrovascular Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tDCS stimulation A (Experimental): Intervention: Transcranial Direct Current Stimulation (tDCS) Up to 20 minutes of tDCS applied to the prefrontal cortex.
  Interventions: Device: Transcranial Direct Current Stimulation
- tDCS stimulation B (Experimental): Intervention: Transcranial Direct Current Stimulation (tDCS) Up to 20 minutes of tDCS applied to the prefrontal cortex.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — TDCS involves sending a weak electrical current to the brain to modulate brain functions.
  Other Names: Neuroelectrics Starstim

SUMMARY:
The purpose of this study is to test the efficacy and safety of tDCS (Transcranial Direct Current Stimulation) on apathy in stroke patients.

DETAILED DESCRIPTION:
Post-stroke apathy is a condition where people show reduced emotions and reduced activity after their stroke, beyond that expected from their degree of weakness. It can occur with, or without, depression, and is associated with more disability and slower recovery. It is thought to be due to dysfunction of the front of the brain (prefrontal cortex). Importantly, there are no proven medical treatments for post-stroke apathy.

Transcranial direct current stimulation (tDCS) is a painless, noninvasive brain stimulation technique that has the potential for alleviating post-stroke apathy. TDCS involves sending a weak electrical current through the head, thereby exciting the brain underneath. This offers potential advantages over medications as tDCS directly targets the brain, while medications need to travel through the bloodstream to reach the brain. TDCS is not an FDA-approved treatment for any condition, but previous trials have shown it may benefit movement and language recovery after stroke, as well as improve thinking ability. Studies have shown tDCS to be very safe with no serious adverse events in over 10,000 subjects studied.

This pilot study will involve three visits to Stony Brook University Hospital. The first is a baseline session where subjects perform all outcome measures but no tDCS is performed other than for familiarization. The second and third sessions are the stimulation sessions where subjects undergo the intervention for 20 minutes to test tDCS effects on the outcome measures. The effects of tDCS for a single session are expected to only last for few hours. Subjects are to receive one type of stimulation in one session and another type in the other session. If this study finds a short term benefit of tDCS for post-stroke apathy it will support a full clinical trial where multiple sessions of tDCS will be given and may provide a long-term benefit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke and radiographically proven ischemic or hemorrhagic stroke (MRI required for ischemic stroke, CT sufficient for hemorrhagic stroke)
* Stroke occurred at least one month prior to first stimulation session
* Ability to provide informed consent
* Availability of a family member / caregiver who knew the subject before the stroke and interacts with the subject on at least a weekly basis
* Score of 6 or higher in initial apathy testing using Apathy Inventory - Clinician score
* Speak English (required for quantifying apathy and performing the cognitive tests)

Exclusion Criteria:

* Other potential cause of apathy including some neurodegenerative diseases, some psychiatric diseases, and anti-dopamine medication
* Prior brain injury (e.g., Traumatic Brain Injury (TBI), stroke) without full motor and cognitive recovery based on patient, family or clinician report
* Active medical illness (e.g., infection, delirium, etc.) that might affect arousal and cognitive function
* Hypoarousal (inability to maintain eye opening without stimulation) from any cause (e.g., stroke, sleep deprivation)
* Any history of epilepsy
* Recent drug or alcohol abuse - within the past year
* Pregnant or breastfeeding
* Moderate to severe aphasia preventing subject from communicating fully
* Any pacemakers, intracranial electrodes, implanted defibrillators, or any other electrical implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Changes in Apathy Inventory Scale - Clinician | at the beginning of each session and 1 day after each session.

SECONDARY OUTCOMES:
Changes in Apathy Inventory Scale - Subject | before and after each stimulation within 2 hours.
Changes in Apathy Inventory Scale - Family/Caregiver | at the beginning of each session and 1 day after each session.
Actimeter | Actimeter is worn from the beginning of the study to end of study (20 to 30 days)
Changes in Language Analysis tests | before and after each stimulation within 2 hours.
Changes in Cognitive Tasks | before and after each stimulation within 2 hours.
Changes in EEG | before and after each stimulation within 2 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Goldfine, MD, Principal Investigator — Stony Brook Medicine
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283